CLINICAL TRIAL: NCT01800175
Title: Non-Significant Risk Feasibility Study to Assess Retention and Replacement of the OTX Punctum Plug
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: OTX-13-001
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation C (Experimental): Two formulations of the OTX Punctum Plug will be evaluated in this trial. The difference in formulations is the time required for degradation of the PEG hydrogel. The persistence of OTX Punctum Plug (Formulation C) is anticipated to be slightly shorter than the persistence of OTX Punctum Plug (Formulation D).
  Interventions: Device: Punctum Plug
- Formulation D (Experimental): Two formulations of the OTX Punctum Plug will be evaluated in this trial. The difference in formulations is the time required for degradation of the PEG hydrogel. The persistence of OTX Punctum Plug (Formulation C) is anticipated to be slightly shorter than the persistence of OTX Punctum Plug (Formulation D).
  Interventions: Device: Punctum Plug

INTERVENTIONS:
Device: Punctum Plug

SUMMARY:
The purpose of this study is to evaluate retention and replacement of the OTX Punctum Plug when placed in the canaliculus of the eyelid. Subjects will be followed for up to 1 year in order to assess retention and replacement of the OTX Punctum Plug for this duration. At the Day 90 visit, subjects will receive a second OTX Punctum Plug after removal of the initial OTX Punctum Plug. The subject will return for visits at Day 180, 270 and 360. On Days 180 and 270, the subject will again receive a new OTX Punctum Plug after the previous OTX Punctum Plug is removed.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be greater than or equal to 40 years of age.
* Subject is in general good health with overall healthy eyes.
* Subject has been informed of the nature of the study and is able to comply with study requirements, the visit schedule and has provided written informed consent, approved by the appropriate IRB.

Exclusion Criteria:

* Presence of any uncontrolled systemic or debilitating disease (e.g. cardiovascular disease, hypertension, diabetes, or cystic fibrosis).
* History of ocular trauma within the past 6 months in either eye.
* History of ocular infection (bacterial, viral, or fungal) or ocular inflammation within 3 months prior to the study in either eye.
* History of chronic or recurrent inflammatory eye disease (i.e., iritis, scleritis, uveitis, herpes keratitis) in either eye.
* History of clinically relevant or progressive retinal diseases such as retinal detachment, retinal degeneration, or diabetic retinopathy in either eye.
* History of any other severe ocular pathology (including severe dry eye) in either eye.
* History of any laser or incisional surgery within 6 weeks prior to the study or scheduled ocular surgery during the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Punctum Plug retention for 90 days post insertion | 360 days
  Retention of the first OTX Punctum Plug through Day 90, retention of the second OTX Punctum Plug through Day 180, retention of the third OTX Punctum Plug through Day 270, retention of the fourth OTX Punctum Plug through Day 360

SECONDARY OUTCOMES:
Successful insertion of a replacement OTX Punctum Plug at Days 90, 180 and 270 | 270 days